CLINICAL TRIAL: NCT05101304
Title: Registre HEAR, Healthcare European Amyloidosis Registry
Status: Recruiting | Type: Observational
Sponsor: Saving Lives Matters (Network)
Responsible Party: Sponsor
Other Study IDs: HR01
Record Dates: First submitted 2021-10-05; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HEAR(Healthcare European Amyloidosis Registry)-Retrospective Cohort: Retrospective collection of deceased patients data with inclusion criteria
- HEAR(Healthcare European Amyloidosis Registry)-Retrospective-Prospective Cohort: Retrospective and prospective collection of patient data and real-life follow-up of patients from the date of inclusion Living patients who met the inclusion criteria
- HEAR(Healthcare European Amyloidosis Registry)-Prospective Cohort: Prospective data collection and real-life follow-up of patients from the date of inclusion These patients are either newly followed in the centre with the inclusion criteria

SUMMARY:
This is a non-interventional, prospective, retrospective, non-comparative, multi-center study.

In order not to interfere with patient management, the study is observational. Thus, no follow-up visit is imposed. The data collection will be limited to the data related to the management of the patients included throughout their follow-up.

This study is intended for all patients with a confirmed or suspected diagnosis of cardiac amyloidosis. Three cohorts will be identified: the HEAR (Healthcare European Amyloidosis Registry)-Retrospective Cohort, the HEAR(Healthcare European Amyloidosis Registry)-Retrospective-Prospective Cohort and the HEAR (Healthcare European Amyloidosis Registry)-Prospective Cohort.

DETAILED DESCRIPTION:
Amyloidosis is a rare disease characterized by infiltration and continuous accumulation of insoluble fibrillar proteins in the extracellular matrix in various organs including kidney, nerve, liver, heart and skeletal muscle. Its prevalence is estimated at 0.5-1.3/100,000. The main forms are:

1. Primary amyloidosis is caused by deposits of monoclonal immunoglobulin light chains produced by a plasma cell clone in the bone marrow.
2. Hereditary (familial) amyloidosis, the major form of which is mutated transthyretin amyloidosis of autosomal dominant transmission. More than 100 different mutations of transthyretin are known and several mutations have been described as amyloidogenic.
3. Systemic senile amyloidosis which is due to deposits of wild-type (unmutated) transthyretin.
4. AA amyloidosis of chronic inflammatory causes.
5. Localized amyloidosis. They are in the vast majority of cases primary amyloidosis (or immunoglobulinic) amyloidosis. The deposition of amyloidosis formed by light chains of antibodies occurs here in contact with a proliferation of plasma cells located in a particular organ. There is no passage of the immunoglobulin light chain into the bloodstream and therefore deposits do not form remotely in other organs.
6. Rare amyloidoses. The prognosis of the disease is most often related to the cardiac involvement. Unfortunately, its diagnosis is often delayed, which worsens the prognosis. This delay is linked to the absence of simple diagnostic tools (biomarkers, imaging, etc.) allowing early diagnosis of the disease. The absence of early diagnostic tools, the heterogeneity of the expression (multi-systemic) of this disease and the difficulty of its management lead to delays in diagnosis and non-management of certain organ disorders, which have an impact on the quality of life of patients.

There is a strong need to help physicians better characterize the clinical and biological presentations of the disease and to improve diagnostic tools and standardize therapeutic management.

All data collected for the study are key, routine data for the condition, readily available in the patients' medical records. It is also possible to use additional and specific computerized tools to collect these data, within the participating expert centers.

Data will be recorded in an electronic observation book.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients must meet all of the following inclusion criteria to be included in the study:

   * Major patient
   * Protected adult patient (guardianship or curatorship)
2. Prospective Cohort:

   Patients referred or who have been referred to the participating centre for suspected amyloidosis.

   Patient who signed the patient information "Prospective Cohort" note
3. Retro-prospective Cohort:

   Patient already followed in the center with a confirmed diagnosis of amyloidosis Patient who signed the "retro-prospective cohort" patient information note
4. Retrospective cohort:

Deceased patients followed in the center with a confirmed diagnosis of amyloidosis

Study participants will not be compensated for their participation

EXCLUSION CRITERIA The patient has expressed his/her refusal to participate Participation in another study, even an interventional one, is not a criterion for non-inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is intended for all patients with a confirmed or suspected diagnosis of cardiac amyloidosis.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The clinical, biological and imaging characteristics of patients with cardiac amyloidosis | 6 years
  Describe the clinical, biological and imaging characteristics of patients with cardiac amyloidosis.

SECONDARY OUTCOMES:
he prevalence and incidence of the different types of amyloidosis and their evolution. | 6 years
  To estimate the prevalence and incidence of the different types of amyloidosis and their evolution.
The therapeutic management (cardiological and specific), their beneficial and secondary effects. | 6 years
  Describe the therapeutic management (cardiological and specific), their beneficial and secondary effects.

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud Pr Damy, Principal Investigator — Henri Mondor University Hospital
Locations (1):
- Hôpital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No